CLINICAL TRIAL: NCT00578760
Title: Does Aspirin Have a Protective Role Against Chemotherapeutically Induced Ototoxicity?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr John Rutka, UNH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Aspirin-01
Record Dates: First submitted 2007-12-18; First posted 2007-12-21 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Hearing Loss; Ototoxicity
Keywords: hearing loss; ototoxicity; cisplatin
MeSH Terms: conditions — Hearing Loss; Ototoxicity | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): placebo OD during course of chemotherapy
  Interventions: Drug: placebo
- 1 (Experimental): 325mg ASA OD during course of chemotherapy
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: aspirin — 325mg ASA OD for the duration of the cisplatin
  Arms: 1
Drug: placebo — OD for course of cisplatin chemotherapy
  Arms: 2

SUMMARY:
Aspirin (ASA) has been shown, in an animal model, to attenuate the ototoxic properties of cisplatin. The researchers plan to investigate this in patients undergoing cisplatin chemotherapy.

The researchers hypothesise that low-dose aspirin can prevent cisplatin induced ototoxicity in the clinical setting.

DETAILED DESCRIPTION:
Cisplatin has the highest ototoxic potential of all platinum containing compounds. It is used in the treatment of squamous cell carcinoma of the head and neck, germ cell tumours of the testis and bladder carcinoma.

42% of 400 patients receiving high-dose cisplatin (70-85 mg/m2, median cumulative dose 420mg) experienced common toxicity criteria (CTC: appendix 1) grade 3 or 4 symptoms (De Jongh 2003). Ototoxicity is dose related: 75-100% of patients receiving a very high dose and 20-40% with a low dose regime will develop significant ototoxic symptoms. In one study, 50% of head and neck cancer patients treated with cisplatin develop ototoxicity (Blakley 1994).

Cisplatin ototoxicity can present as a variable collection of symptoms and signs. These include bilateral and symmetrical hearing loss that is permanent and irreversible. High frequency sensorineural hearing loss with progression towards lower frequencies. Tinnitus, that is also permanent and irreversible.

There are a number of known factors that can predispose to cisplatin ototoxicity. They include: Dose, duration and mode of administration, age extremes, previous or concurrent cranial irradiation, previous history of hearing loss, renal disease, concomitant use of other ototoxic drugs, noise exposure with concomitant cisplatin administration, decreased serum albumin level, low hemoglobin level, low red blood cell count and a low haematocrit. Interestingly, cisplatin ototoxicity is considered to be exclusively confined to the cochlear, the vestibular system is unaffected (Myers 1993).

Ototoxicity from chemotherapeutic agents is due, in part, to reactive oxygen species. Reactive oxygen species can be attenuated by antioxidants. Salicylates are antioxidants that can be administered as aspirin.

It has been shown, in an animal model, that aspirin can protect hearing from cisplatin induced ototoxicity (Li 2002). In this set of experiments, the rat was used to evaluate the protective role of aspirin in both the acute and chronic setting. Auditory evoked brain stem responses were used to determine pre- and post-intervention hearing thresholds. In the acute experiments (n=23), one dose of cisplatin (16mg/kg) was administered and the animals were given aspirin (100mg/kg) starting the day before cisplatin treatment and continuing 4 days thereafter. There was a significant difference in hearing thresholds between the treatment and control groups at 3, 8 and 14kHz.

In the chronic experiments cisplatin was given on days 1, 4 and 7 (5mg/kg). Aspirin was given from 2 days before to 3 days after cisplatin treatment (100mg/kg bd). The hearing thresholds were compared before the first dose and 10 days after the last treatment. In those animals treated concurrently with aspirin, their hearing did not differ form control animals at 16 and 24 kHz. This was correlated to a significant reduction in inner hair cell loss from 20% (cisplatin) to 8% (cisplatin and aspirin).

Salicylates also protected renal function as determined by both plasma blood urea nitrogen and creatinine levels.

Salicylates did not affect tumour mass or metastasis. The rats were inoculated with malignant breast cancer cells (metastatic mammary adenocarcinoma). Aspirin protected against cisplatin-induced ototoxicity, without affecting the oncolytic action of the cisplatin.

Gentamicin and cisplatin both have a similar ototoxic mechanism of action. Aspirin has been shown to prevent gentamicin-induced hearing loss without compromising its anti-bacterial efficacy in both animal models and the clinical setting (Sha 2006, Chen 2007). Sha's group reported a prospective, randomized, double-blind trial with 200 patients. The patients all required gentamycin for clinical indications. In the 'treatment' arm of the study, the patients also received aspirin (1g tds for 14 days). A significant difference in hearing was shown at 6 and 8kHz of >15dB if aspirin was not given.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cisplatin treatment for the following malignancies:

  * germ-cell
  * bladder
  * head and neck (Only head and neck patients requiring only 2 cycles of post-operative chemo-radiotherapy, and therefore not requiring a gastrostomy tube, will be enrolled.)
* Over 18 years of age
* Normal otoscopic examination
* Informed consent

Exclusion Criteria:

Patients with the following will be excluded:

* Not able to grasp the study implications or unable to consent.
* History of peptic ulcer disease
* Severe renal impairment (U&E, Cr clearance)
* Haemophilia
* Severe hepatic impairment
* Cerebrovascular haemorrhage
* Acute gout
* Hypersensitivity to NSAIDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2008-02; Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
hearing loss | before and after chemotherapy

SECONDARY OUTCOMES:
hearing loss and tinnitus questionnaires | before and after cisplatin treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada